CLINICAL TRIAL: NCT03754361
Title: The Study of Efficacy and Safety of Automated Peritoneal Dialysis in Urgent Start Dialysis as Compared With Intermittent Hemodialysis in ESRD Patients,a Multi-center, Non-blind and Controlled Clinical Trial
Brief Title: The Study of Efficacy and Safety of Automated PD in Urgent Start Dialysis
Acronym: URG-APD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient recruitment difficulties
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: First Hospital of China Medical University (Other); Beijing Anzhen Hospital (Other); The Luhe Teaching Hospital of the Capital Medical University (Other); Ningbo No.2 Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URG-APD
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-09

CONDITIONS: ESRD
Keywords: urgent start dialysis; automated PD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: the mode of urgent dialysis will choose by patient guided by nephrologist, the HD group will receive the standard traditional treatment: from induction HD to regular HD. The PD group will receive the APD daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APD group (Experimental): Subjects will receive PD catheter placement and subsequent automated peritoneal dialysis treatment
  Interventions: Procedure: automated peritoneal dialysis
- IHD group (Active Comparator): Subjects will receive un-tunneled hemodialysis catheter placement and subsequent hemodialysis treatment 3-4 times per week,2-4 hours each time.
  Interventions: Procedure: IHD

INTERVENTIONS:
Procedure: automated peritoneal dialysis — peritoneal dialysis administered by a cycler
  Arms: APD group
Procedure: IHD — HD 4hour 2-3times per week
  Arms: IHD group

SUMMARY:
This is a multi-center, controlled clinical trial study. The purpose of this study is to examine the efficacy and safety of automated peritoneal dialysis as compared with intermittent haemodialysis for ESRD patients with indications for urgent start dialysis.

DETAILED DESCRIPTION:
Hemodialysis（HD） and peritoneal dialysis (PD) are both the main methods to treat with end-stage renal disease (ESRD) uremia patients. The first 3-month mortality and hospitalization rate of new dialysis patient is much higher than that of regular dialysis's. So it is very important to set up dialysis pathway and from inducing dialysis into regular dialysis smoothly. But in the global 50-70%, more than 70% of the patients in China can not establish the dialysis pathway in advance according to the plan. With the common, a temporary deep venous catheter would be used first, then the fistula established later, as the final transition for hemodialysis. Urgent peritoneal dialysis can be established 24 hours after the establishment of permanent access dialysis, simply and easily, it can protect the residual kidney function; reduce treatment costs, hemodynamic stability, no anticoagulant is its unique advantages, At the same time, also avoid the temporary deep venous pathway prone to local bleeding, infection, venous thrombosis, central venous stenosis, direct impact on the future of the mature of fistula , or transplanted kidney vascular conditions. Automatic peritoneal dialysis (APD) in the treatment of urgent dialysis patients can save more manpower and resources, and improve the efficiency of peritoneal dialysis. The study on the efficacy and safety of urgent dialysis lacks the precisely designed multi-center, prospective and controlled clinical trial, and APD only induces 3 days, it is difficult to really reflect the safety and effectiveness of APD. Therefore, it is of great practical significance to study the difference of safety, efficacy and cost-effectiveness between urgent PD and HD in a prospective, control and multicenter clinical trial. 206 ESRD uremia patients will involve in this multi-center, prospective and controlled clinical trial, the mode of urgent dialysis will choose by patient guided by nephrologist, the HD group will receive the standard traditional treatment: from induction HD to regular HD. The PD group will receive the APD daily. All patient will be monitor the physiological and biochemical marker for 14 day, and all adverse events and dead within 90days will collected to evaluated the safety, efficacy of the two urgent dialysis modes.

ELIGIBILITY:
Inclusion Criteria:

* CKD(chronic kidney disease)-5 stage patient whose eGFR（CKD-EPI（chronic kidney disease-epidemiology collaboration））<15 ml/min/1.73m2,occured uremic symptoms or volume overload need of renal replacement therapy(RRT) within 14 days .
* Prolonged RRT access is not available.
* No dialysis treatment was given within 1 months.
* The vital signs are stable and tolerable in peritoneal dialysis catheterization or central venous catheterization.
* Able to understand the whole process of the trial, voluntarily participate in and sign informed consent.

Exclusion Criteria:

* Maintenance RRT alraedy.
* Serious metabolic disorders ( hyperkalemia and acidosis) cause significant changes in electrocardiogram or other emergency indications to RRT within 24 hours.
* Hypertensive emergencies(diastolic blood pressure>130mmHg)
* Severe respiratory, circulatory or hepatic failure requires instrumental support or vasoactive drugs to maintain vital signs.
* High catabolic state eg. severe inflammation or trauma
* Absolute contraindication of peritoneal dialysis such as recent abdominal surgery (<1month), multiple abdominal surgeries.
* Absolute contraindication for hemodialysis such as hemodynamic instability (systolic blood pressure <80mmHg).
* Pregnant.
* Expected to survive for less than 1 years.
* Plan for kidney transplantation within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
infective morbidity | At 14 days after the initiation of dialysis
  peritonitis (APD), Bacteremia and catheter-related infections (APD and IHD)

SECONDARY OUTCOMES:
Mechanical complications morbidity | At 14 and 90 days after the initiation of dialysis
  catheter leakage and migration (APD), catheter obstruction (IHD)， Exit site bleeding, pneumothorax, hernia
dialysis related mortality | At 14 and 90 days after the initiation of dialysis
  catheter-related:Sepsis, severe thromboembolic events (massive cerebral infarction, pulmonary embolism), arrhythmia (ventricular tachycardia, ventricular fibrillation),bleeding, Congestive heart failure and ischemic heart disease
infective morbidity | At 90 days after the initiation of dialysis
  peritonitis (APD), Bacteremia and catheter-related infections (APD and IHD)

CONTACTS AND LOCATIONS:
Overall Officials: Limeng Chen, MD, Principal Investigator — Division of Nephrology, Peking Union Medical College Hospital
Locations (5):
- China (5):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Ningbo No.2 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
To comply with laws in China, local regulations and hospital policy, IPD sharing might be restricted